CLINICAL TRIAL: NCT00509080
Title: Prognosis in Asymptomatic Mitral Regurgitation (PAMIR) Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Schweizerische Herzstiftung (Other)
Responsible Party: Sponsor
Other Study IDs: PAMIR
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Mitral Regurgitation
Keywords: mitral regurgitation; BNP; NT-proBNP; natriuretic peptides; valvular heart disease
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine if the use of BNP/NT-proBNP levels in the detection of early left ventricular dysfunction and damage may improve the timing of cardiac surgery and therefore the long-term management of asymptomatic patients with severe mitral regurgitation.

DETAILED DESCRIPTION:
Background: One of the most difficult issues in the care of asymptomatic patients with severe valvular heart disease, particularly mitral regurgitation, is the timing of the surgical intervention. Unlike the stenotic lesions, regurgitant lesions often progress insidiously, causing left ventricular damage before symptoms develop. Current criteria for surgical intervention include left ventricular dimensions and left ventricular ejection fraction. The clinical problem is that once these morphologic criteria are fulfilled, the prognosis has already worsened, even if surgery is performed promptly. In addition, the onset of symptoms may be difficult to detect because of physical inactivity or under-reporting. In some patients, it may be unclear whether symptoms are related to valvular heart disease or other conditions.

Natriuretic peptides including B-type natriuretic peptide (BNP) and NT-proBNP may be more sensitive markers of left ventricular damage than morphologic studies such as echocardiography. The use of BNP or NT-proBNP levels may help timing the surgical intervention before irreversible left ventricular damage has occurred. Previous experience with BNP and NT-proBNP testing in patients with valvular heart disease is limited, albeit promising.

Aim: To test the hypotheses that:

* Elevated BNP/NT-proBNP levels reflect early left and right ventricular dysfunction indicating imminent congestive heart failure and cardiac decompensation, and call for surgical intervention.
* The BNP/NT-proBNP level is a more sensitive marker of ventricular damage than ventricular dimensions and left ventricular ejection fraction.
* Low BNP/NT-proBNP levels indicate a low event rate with medical therapy and may therefore reassure a "wait and see strategy".

Patients and methods: The prospective cohort study is designed to enrol 200 patients with severe mitral regurgitation and followed over a 4-year period. Natriuretic peptides including BNP and NT-proBNP will be measured in addition to detailed clinical, electrocardiographic, and echocardiographic assessment prospectively and repetitively in patients with severe mitral regurgitation during routine consultations at 6 months intervals. Our primary analysis (longitudinal study) will focus on the prognosis in asymptomatic patients. In addition, a sub-study will also include symptomatic patients with severe mitral regurgitation whether or not they are scheduled to undergo valvular surgery (cross sectional study) in order to obtain more reliable data regarding BNP/NT-proBNP levels in patients with a formal indication for valvular surgery. The treating physician will remain blinded to the BNP/NT-proBNP values. In this cohort study, we will try to identify a BNP/NT-proBNP cut-off values that predict major adverse cardiac events including cardiac death, congestive heart failure, myocardial infarction, or persistent left ventricular systolic dysfunction at 6 months after valvular surgery.

Clinical Significance: The use of BNP/NT-proBNP levels in the detection of early left ventricular dysfunction and damage may improve the timing of cardiac surgery and therefore the long-term management of asymptomatic patients with severe mitral regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe isolated mitral regurgitation due to valvular disease

Exclusion Criteria:

* Missing written patient consent
* Active infective endocarditis
* Relative mitral regurgitation due to left ventricular disease
* Other moderate to severe dysfunctional valve
* Previous cardiac surgery
* Pregnancy
* Sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Composite of congestive heart failure, decompensated heart failure and valve surgery | 360 days
  Elevated BNP/NT-proBNP levels reflect early left and right ventricular dysfunction indicating imminent congestive heart failure and cardiac decompensation, and call for surgical intervention.
Composite of congestive heart failure, decompensated heart failure and valve surgery | 720 days
  Elevated BNP/NT-proBNP levels reflect early left and right ventricular dysfunction indicating imminent congestive heart failure and cardiac decompensation, and call for surgical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Mueller, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (6):
- Germany (3):
  - Herz-Zentrum Bad Krozingen, Bad Krozingen
  - Kerkhoff Klinik, Bad Nauheim
  - Cardiology Praxis Dr. Gekeler, Loerrach
- Switzerland (3):
  - Cardiology Praxis Dr. Cron/ Dr. Hess, Basel
  - Cardiology Praxis Prof. A. Hoffmann, Basel
  - University Hospital of Basel, Basel

IPD SHARING:
Plan to Share IPD: No